CLINICAL TRIAL: NCT01744080
Title: Effect of Surgical Wait Times on Outcomes of Rotator Cuff Surgery
Brief Title: Rotator Cuff Injury to Surgery
Acronym: RC-IS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistic issues could not be resolved - study closed without any patients recruited
Sponsor: Panam Clinic (Other)
Responsible Party: Principal Investigator, Peter MacDonald, Department Head, Orthopaedics, Panam Clinic
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2012:112
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Rotator Cuff Tear
Keywords: Rotator cuff
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Surgery (Active Comparator)
  Interventions: Other: Early Surgery
- Regular Wait Time (Experimental)
  Interventions: Other: Regular Wait Time

INTERVENTIONS:
Other: Regular Wait Time — Surgery will take place no earlier than 9 months and no later than 12 months after the sport medicine physician consult.
  Arms: Regular Wait Time
Other: Early Surgery — Patient will proceed to have rotator cuff repair surgery within 3 months of the initial consult with the sport medicine physician.
  Arms: Early Surgery

SUMMARY:
The purpose of this prospective randomized controlled trial is to compare post-operative outcome between participants undergoing expedited surgery compared to those proceeding through a 'typical' wait time process. A secondary purpose is to evaluate the progression of rotator cuff tear size from the time of initial consult to the time of surgery.

DETAILED DESCRIPTION:
Consented patients will undergo a pre-operative assessment conducted by a study physiotherapist, including the following: 1) demographic information (age, gender, height, weight, smoking status, employment, recreational activities, time of injury, etc.); 2) shoulder ROM, 3) shoulder strength using a handheld dynamometer, and 4) subjective shoulder-specific outcome measures which include the Western Ontario Rotator Cuff Score (WORC), American Shoulder and Elbow Score (ASES), and Simple Shoulder Test (SST). Measurement of tear size will also be documented by an experienced radiologist from the initial MRI or ultrasound.

Patients will undergo initial consultation with the orthopaedic surgeon to confirm suitability for surgical management. If deemed appropriate to continue as a participant, the individual participants will be randomized to one of the two study groups. If in the Expedited group, the patient will proceed to have rotator cuff repair surgery within 3 months of the initial consult with the sports medicine physician. If randomized to the Control or 'Typical Wait Time' Group, surgery will take place no earlier than 9 months and no later than 12 months after the sports medicine physician consult.

Just prior to surgery, a second diagnostic imaging test will take place, either ultrasound or MRI, to document progress in tear size and any secondary pathology in the control group. Diagnostic test findings will be confirmed intraoperatively. All rotator cuff repairs will be performed by one of four fellowship trained orthopaedic surgeons.

The control study group will be sent the subjective questionnaires at 8 week intervals while they are waiting for surgery. Post-surgery study follow-ups will take place at 6, 12, and 24 months for both groups. All patients will be provided with the same rehabilitation protocol including pain management, range of motion and strengthening exercises. The same data as that collected pre-surgery will be repeated as well as any occurrences of failure of the repair. Failure of the repair is defined as ongoing severe pain, limited ROM, and/or decreased strength. If a failure occurs, follow-ups will continue until 24 months following failure or 24 months following revision surgery, if performed.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 45 and 70 years old
* Acute full-thickness rotator cuff tear of supraspinatus an/or infraspinatus (as confirmed by appropriate diagnostic imagine)

Exclusion Criteria:

* Presence of a tear of the subscapularis and/or teres minor;
* Presence of a partial-thickness tear of the supraspinatus/infraspinatus;
* Patient has undergone previous RC surgery to the affected shoulder;
* Patient has an active WCB Claim or prior claim related to their shoulder;
* Previous major joint trauma, infection, or avascular necrosis;
* Chronic dislocation, inflammation, or degenerative glenohumeral arthropathy;
* Evidence of significant cuff arthropathy (superior glenohumeral translation and/or acromial erosion, as diagnosed by diagnostic imaging)
* Psychiatric illness, cognitive impairment, or other health condition (i.e. visual impairment) which precludes informed consent or renders the patient unable to complete study questionnaires
* Major medical illness where life expectancy is less than 2 years;
* Does not speak/read/understand English;
* No fixed address or means of contact;
* Unwillingness to complete necessary follow-ups

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2017-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Western Ontario Rotator Cuff | 24 months
  WORC score questionnaire is a tool designed for self-assessment of shoulder function for patients with rotator cuff problems. Difference between study arm outcomes will be assessed using pre-op WOSI score as a covariate

SECONDARY OUTCOMES:
American Shoulder and Elbow Surgeons (ASES) | 24 months
  The ASES assessment (patient report section) is a region-specific questionnaire designed for self-assessment of aspects of pain and function. Difference between study arm outcomes will be assessed using pre-op ASES score as a covariate

OTHER OUTCOMES:
Injury to Surgery Time | 24 months
  Time will be calculated from initial injury to consultation to surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Leiter, MSc, PhD, Principal Investigator — Pan Am Clinic
Locations (1):
- Pan Am Clinic, Winnipeg, Manitoba, Canada